CLINICAL TRIAL: NCT03974191
Title: 13-year Follow-up of Women With Chronic Low Back Pain in Primary Care - a Prospective Longitudinal Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: VGFOUREG855601
Record Dates: First submitted 2019-05-27; First posted 2019-06-04 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Low Back Pain; Chronic Widespread Pain; Predictors; Pain; Physical Activity; Work Ability
Keywords: Low Back Pain; Pain; Physical Activity; Physical Capacity; Work Ability; Primary Health Care
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Pain; Motor Activity | interventions — Functional Status; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 131 participants with chronic low back pain: All the participants (n=131) with chronic low back pain (CLBP) from the cross-sectional study in 2006 are invited to participate in the present 13-year follow-up. The same examination battery used in the cross-sectional study plus a supplementary Chair Stand Test will be used.
  Interventions: Other: Change in function, activity, participation and other health related factors in CLBP and to identify predictors for pain, activity and work ability after 13 years.

INTERVENTIONS:
Other: Change in function, activity, participation and other health related factors in CLBP and to identify predictors for pain, activity and work ability after 13 years. — 13-year prospective longitudinal cohort study

SUMMARY:
Background: Low back pain (LBP) is among the main causes of long-term sickness absence and is associated with considerable costs for both the individual and society. LBP affects 60-80% of the population and most individuals recover, while about 10-20% develop persistent pain and disability. Women have a higher risk of developing chronic LBP (CLBP) and widespread pain.

Purpose: To investigate change in body function, activity, participation and other health related factors in women with CLBP after 13 years and to identify prognostic factors for pain, activity limitation and work ability.

Methods: In the present study, all women (n = 131) who were included in the cross-sectional study in 2006 and who were followed-up after 2 years are now invited to the same study-protocol 13 years after the first examination in 2006.

The Swedish Ethical Review Authority approved the study. Dnr: 2019-01944, 2019-05-21.

DETAILED DESCRIPTION:
Background: Low back pain (LBP) is among the main causes of long-term sickness absence and is associated with considerable costs for both the individual and society. LBP affects 60-80% of the population and most individuals recover, while about 10-20% develop persistent pain and disability. Women have a higher risk of developing chronic LBP (CLBP) and widespread pain.

How LBP develops into recurrent and or more persistent pain with disability is not fully understood. Prognostic factors for pain development, work ability and self-rated activity limitation in 1 and 2-year follow-ups of persons with CLBP who sought primary care are described. Performance on physical capacity tests (6-min walking test), limitations on self-rated activity and participation and psycho-social factors play a role in unfavorable pain and function development. However, there are patients with CLBP who have no anatomical, demographic or psychosocial explanation of their symptoms. Some people with CLBP also have widespread pain and show altered pain sensitivity as fibromyalgia.

Purpose:To investigate change in body function, activity, participation and other health related factors in women with CLBP after 13 years and to identify prognostic factors for pain, activity limitation and work ability.

Methods: In the present study, all women (n = 131) who were included in the cross-sectional study in 2006 and who were followed-up after 2 years are now invited to the same study-protocol 13 years after the first examination in 2006.

Participants will be assessed by a registered physiotherapist at one occasion. Demographic data are collected, Questions about social support, sleep quality and sleep quantity, smoking and alcohol consumption. Self-reported questionnaires, pain and function performance tests will be assessed.

Data Analysis: Descriptive analysis based on data level; mean value (standard deviation), median (25th; 75th percentile), number and proportion will be used to present the group's characteristics. For analysis of change between the first assessment and after 13 years, Wilcoxon's signed rank test will be used for continuous variables and Teckentest / McNemar's test will be used for nominal data.

Multivariable regression analysis will be performed to calculate predictors of pain intensity (VAS), number of pain locations/pain distribution, self-rated activity limitation (RMDQ) and work ability after 13 years. Independent variables will be variables at the first assessment within the domains; body function (pain intensity, pain distribution, pain sensitivity, anxiety, depression, function test and stress), activity (RMDQ) and participation (work ability), as well as other health-related factors (Health-Related Quality of Life (SF-36), Leisure Time Physical Activity Instrument, Experience of Physical Activity). Multivariable regression models will be adjusted for age, level of education and social status. P-value is set to 0.05.

Ethical approval: The Swedish Ethical Review Authority approved the study. Dnr: 2019-01944, 2019-05-21.

Expected Results: The results is expected to provide knowledge about long-term clinical course (13 years) and prognostic factors for a positive pain and function development of CLBP in women seeking primary care.

ELIGIBILITY:
Inclusion Criteria:

* All participants (n=131) included in the Cross Sectional Study in 2006

Exclusion Criteria:

* Pregnant
* Serious somatic disorders
* Serious psychiatric disorders

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study will follow up all women (n=131) included in the cross sectional study in 2006.
Study Population: The 183 women who fulfilled the inclusion criteria were invited to participate in the cross-sectional study in 2006 and 131 accepted participation. All 131 from the cross-sectional study are now invited to participate in the present 13-year follow-up.The inclusion criteria at the first assessment in 2006 were: female patient, age between 18 and 60 years, low back pain (pain between costal margins and gluteal folds) with or without referred leg pain. Further criteria were; greater than 12-week's duration of symptoms, not pregnant, no known spinal disorders, no other severe somatic or psychiatric disorders, understanding in Swedish.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Activity limitation | 2019, change from the first assessment (2006) to the present 13-year follow-up (2019), identify predictors (2006) for activity limitation (RMDQ) at the 13-year follow-up
  Roland and Morris Disability Questionnaire (RMDQ) will be used.
Pain intensity | 2019, Change from the first assessment (2006) to the present 13-year follow-up (2019), identify predictors (2006) for pain intensity (VAS) at the 13-year follow-up.
  A Visual Analogue Scale (VAS), ranging 0 to 100 mm will be used for pain intensity during the last week. 0 mm indicates no pain and 100 mm indicates very severe pain. Higher score indicates more severe pain.
Work ability | 2019, Comparison from the first assessment (2006) to the present 13-year follow-up (2019), identify predictors (2006) for work ability at the 13-year follow-up.
  Sick-leave periods, and sickness and activity compensation is obtained from the Swedish Social Insurance Agency's MiDAS database. Self-reported work status dichotomized into two categories, work ability or not will be used.

SECONDARY OUTCOMES:
Pain distribution | 2019, Comparison from the first assessment (2006) to the present 13-year follow-up (2019), identify predictors (2006) for pain distribution at the 13-year follow-up.
  A drawing of the body will be used for assessing distribution of pain

OTHER OUTCOMES:
Walking capacity | 2019, Change from the first assessment (2006) to the present 13-year follow-up (2019).
  The 6-minute walk test (6MWT) will be used. The person walks back and forth in a measured distance of 30 meters for 6 minutes. The number of meters achieved is recorded.
Lower limb muscle endurance and muscle strength | 2019
  The Chair Stand Test (CST) will be used.
Hand grip strength | 2019, Change from the first assessment (2006) to the present 13-year follow-up (2019).
  The Grippit®, electronic hand strength measurement will be used. Sustained hand grip strength will be measured during 10 seconds for each hand.
Hand grip strength | 2019
  The Jamar Hand Dynamometer®, will be used for measuring hand grip strength for each hand.
Pain sensitivity/pain threshold | 2019, Change from the first assessment (2006) to the present 13-year follow-up (2019).
  Somedic algometer® will be used.
Fatigue | 2019, Change from the first assessment (2006) to the present 13-year follow-up (2019).
  Multidimensional Fatigue Inventory (MFI-20) will be used.
General fatigue | 2019, Change from the first assessment (2006) to the present 13-year follow-up (2019).
  A Visual Analogue Scale (VAS), ranging 0 to 100 mm will be used for general fatigue during the last week. 0 mm indicates no tiredness and 100 mm indicates very tired. Higher score indicates more severe general fatigue.
Sleep quantity | 2019, Change from the first assessment (2006) to the present 13-year follow-up (2019).
  One question will be used: "Do you think you get enough sleep?" (Range 1-4). Higher score indicate better sleep quantity.
Sleep quality | Time frame: 2019, Change from the first assessment (2006) to the present 13-year follow-up (2019)
  One questions will be used: "On the whole, how do you think you sleep?" (Range 1-4). Higher score indicate better sleep quality.
Social support | 2019, Change from the first assessment (2006) to the present 13-year follow-up (2019).
  The 4-item version of Medical Outcome Study Social Support Survey will be used.
Stress | 2019, Change from the first assessment (2006) to the present 13-year follow-up (2019).
  Stress and Crisis Inventory (SCI-93) will be used for measuring clinical symptoms of stress.
Physical function | 2019, Comparison from the first assessment (2006) to the present 13-year follow-up (2019).
  The Patient Specific Functional Scale (PSFS), will be used for the participant´s self-identified activities that are difficult to perform due to low back pain. Then the participant rates the level of difficulty for each identified activity on an 11-point numeric scale ranging from 0 ("unable to perform activity") to 10 ("able to perform activity unhindered or at pre-injury level").
Leisure Time Physical Activity | 2019, Change from the first assessment (2006) to the present 13-year follow-up (2019).
  Leisure Time Physical Activity Instrument (LTPAI) will be used to assess the amount of self-rated physical activity in free time during a typical week
Experience of physical activity | 2019, Change from the first assessment (2006) to the present 13-year follow-up (2019).
  Experience of physical activity questionnaire will be used.
Risk for long-term disability and sick-leave | 2019, Change from the first assessment (2006) to the present 13-year follow-up (2019).
  Örebro Musculoskeletal Pain Screening Questionnaire (ÖMPSQ), estimate the risk for long-term disability and sick-leave. The sum score of 21 items will be used.
Health-related quality of life | Change from the first assessment (2006) to the present 13-year follow-up (2019).
  Short Form-36 (SF-36) will be used to measure health-related quality of life.
Alcohol consumption | Comparison from the first assessment (2006) to the present 13-year follow-up (2019).
  The Alcohol Use Disorders Identification Test (Audit-C) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Nordeman, PhD, Principal Investigator — R&D primary care Region Västra Götaland, University of Gothenburg Sweden
Locations (3):
- Sweden (3):
  - Närhälsan, Region Västra Götaland, Alingsås
  - R&D primary care, Region Västra Götaland, Borås
  - Närhälsan, Region Västra Götaland, Uddevalla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nordeman L, Gunnarsson R, Mannerkorpi K. Prevalence and characteristics of widespread pain in female primary health care patients with chronic low back pain. Clin J Pain. 2012 Jan;28(1):65-72. doi: 10.1097/AJP.0b013e318223622c. PMID 21677567